CLINICAL TRIAL: NCT07029503
Title: Swedish Cardiac And Renal Failure Study-1 (SCARF-1): An Open-Label Pilot Trial to Evaluate the Feasibility, Safety and Efficacy of Eplerenone in Patients With Heart Failure With Reduced Ejection Fraction and Severe Chronic Kidney Disease
Brief Title: Swedish Cardiac And Renal Failure Study-1
Acronym: SCARF-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Carl Haggård, MD, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCARF-1; 2025-520550-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-02; First posted 2025-06-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HFrEF - Heart Failure With Reduced Ejection Fraction; Chronic Kidney Disease
Keywords: HFrEF - Heart Failure with Reduced Ejection Fraction; Chronic kidney disease; Heart failure; Chronic heart failure; HFrEF; CKD; Renal dysfunction; Kidney dysfunction; Renal impairment; Advanced; Severe; Mineralocorticoid receptor antagonists; MRA; Eplerenone; Sodium Zirconium Cyclosilicate; SZC
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure; Renal Insufficiency; Lymphoma, Follicular | interventions — Eplerenone

STUDY DESIGN:
Intervention Model Description: ABA-design with a 12-week baseline, a 12-week intervention, and a 12-week withdrawal period. Two observational periods are chosen due to the high risk of natural clinical deterioration, even over a relatively short timeframe, and to enable within-participant comparison of outcome slopes across phases.
Masking Description: Transthoracic Echocardiography (TTE) analysis will take place retrospectively in a blinded manner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Experimental): Eplerenone
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Participants will receive eplerenone 25 mg once daily or every other day, based on baseline potassium levels, eGFR, systolic blood pressure, and concomitant use of weak or moderate CYP3A4 inhibitors.
  The study will implement a safety protocol with predefined procedures for managing significant hyperkalemia, worsening renal function, and hypotension. These will include temporary or permanent dose reduction or discontinuation of eplerenone, and, if necessary, administration of the potassium binder sodium zirconium cyclosilicate (SZC, Lokelma®).
  Other Names: Inspra®

SUMMARY:
Previous studies have shown that patients with heart failure with reduced pumping function and preserved kidney function experience improved symptoms, longer survival, and fewer hospitalizations when treated with medications such as eplerenone. However, individuals with impaired kidney function have been excluded from these trials due to concerns about potential adverse effects on potassium levels, kidney function, and possibly also blood pressure. As a result, clear treatment recommendations for this high-risk group are lacking.

In recent years, however, background therapies have been modernized and are now associated with a lower risk of potassium disturbances. Preliminary data also suggest that patients with impaired kidney function may benefit from eplerenone treatment. However, confirmation through dedicated studies is needed.

The primary objective of this pilot trial is to assess the feasibility and safety of eplerenone in patients with heart failure with reduced pumping function and impaired kidney function. Treatment effectiveness will also be explored.

DETAILED DESCRIPTION:
Virtually all major trials in heart failure with reduced ejection fraction (HFrEF), including those investigating mineralocorticoid receptor antagonists (MRAs) such as eplerenone, have excluded patients with severe chronic kidney disease (CKD). This exclusion has likely been driven by concerns over the risks of hyperkalemia and worsening renal function (WRF). However, post-hoc analyses of these major trials, along with data from registries and cohort studies, suggest that patients with more advanced renal impairment may still derive an overall benefit from MRA treatment.

The objective of this pilot trial is to evaluate the feasibility and safety of eplerenone in patients with HFrEF and severe CKD. An exploratory analysis of efficacy will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* The participant has given their written consent to participate
* A diagnosis of HFrEF according to current criteria, for at least three months before the screening visit
* Echocardiography within 24 months of the screening visit with ejection fraction ≤ 40%. The responsible investigator is allowed to order a new TTE at their own discretion if clinically indicated - e.g. following the initiation of markedly intensified HFrEF-treatment or in the event of significant clinical deterioration. If the new TTE shows an EF > 40%, the participant will not be eligible for inclusion. However, a potential echocardiographic worsening should not, by itself, preclude enrollment
* New York Heart Association class II-III
* Optimally treated and stable HFrEF (according to the investigator) since at least four weeks before the screening visit. Treatment should include beta-blockers, sodium/glucose co-transporter 2 inhibitors, angiotensin-converting enzyme inhibitors, or angiotensin receptor blockers if eGFR ≥ 20 ml/min/1.73m2 according to the revised Lund-Malmö method. Participants should also have cardiac resynchronization therapy or an implantable cardioverter-defibrillator if the indication exists according to current guidelines
* eGFR < 30 ml/min/1.73m2 according to the revised Lund-Malmö method at least once during the 12 months before the screening visit, and eGFR < 45 ml/min/1.73m2 at the time of inclusion

Exclusion Criteria:

* P-K ≥ 5.6
* For the first ten study participants:

eGFR < 20 ml/min/1.73m2 according to the revised Lund-Malmö method, or projected decline in eGFR to < 10 ml/min/1.73m2 during the 36-week study period. The projected decline will be estimated using the three most recent eGFR values from the previous 6-12 months

- For the remainder of the study participants: eGFR < 10 ml/min/1.73m2 according to the revised Lund-Malmö method, or projected decline in eGFR to < 10 ml/min/1.73m2 during the 36-week study period. The projected decline will be estimated using the three most recent eGFR values from the previous 6-12 months

* Ongoing/planned dialysis
* Systolic blood pressure < 90 mmHg
* Uncontrolled hypertension as judged by the investigator
* Severe hepatic impairment (Child-Pugh C)
* History of, or planned, heart transplantation or left ventricular assist device
* Unwillingness to comply with highly effective contraceptive methods, or ongoing/planned pregnancy, or breastfeeding
* Previous allergic reaction to an MRA or a potassium binder
* Ongoing treatment with lithium, cyclosporine, tacrolimus, nonsteroidal anti-inflammatory drugs, trimethoprim, or strong CYP3A inhibitors (ketoconazole, itraconazole, ritonavir, nelfinavir, clarithromycin, telithromycin, and nefazodone) or inducers (rifampicin, carbamazepine, phenytoin, phenobarbital, and St. John's Wort)
* QTc(f) ≥ 550 msec, history of QT prolongation associated with any medication requiring medication discontinuation, or congenital long QT syndrome
* Uncontrolled arrhythmia as judged by the investigator
* Acute cardiac hospitalization or procedure within four weeks before inclusion
* Not suitable as judged by the investigator (presumed inability to participate, severe or terminal co-morbidity, and expected survival < 12 months)
* Previously enrolled in this trial or participation in another trial not approved for co-enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of participants who complete the treatment period with and without the need to use a potassium binder | Between the first and final day of the 12-week eplerenone treatment period
  Without eplerenone interruption/discontinuation due to safety reasons, with and without SZC

SECONDARY OUTCOMES:
The occurrence of plasma potassium (P-K) ≥ 5.6 and ≥ 6.0 | Between the first and final day of each of the three 12-week study periods
  Yes/no
Hospitalization for hyperkalemia | Between the first and final day of each of the three 12-week study periods
  Primary or co-primary reason, yes/no
The occurrence of P-K < 3.0 | Between the first and final day of each of the three 12-week study periods
  Yes/no
Hospitalization for hypokalemia | Between the first and final day of each of the three 12-week study periods
  Primary or co-primary reason, yes/no
Decrease in eGFR of ≥ 30% and ≥ 50% | Between the first and final day of each of the three 12-week study periods
  According to the revised Lund-Malmö method in ml/min/1.73 m2, compared to the start of each study period, yes/no
Hospitalization for renal failure | Between the first and final day of each of the three 12-week study periods
  Primary or co-primary reason, yes/no
Initiation of dialysis | Between the first and final day of each of the three 12-week study periods
  Yes/no
Participant-reported lightheadedness due to orthostatic hypotension as judged by the investigator | Between the first and final day of each of the three 12-week study periods
  Yes/no
Participant-reported syncope | Between the first and final day of each of the three 12-week study periods
  Yes/no
Any participant-reported side effect | Between the first and final day of each of the three 12-week study periods
  Yes/No
Hospitalization for heart failure | Between the first and final day of each of the three 12-week study periods
  Primary or co-primary reason, yes/no
All-cause hospitalization | Between the first and final day of each of the three 12-week study periods
  Yes/no
Cardiovascular death | Between the first and final day of each of the three 12-week study periods
  Primary reason, yes/no
All-cause death | Between the first and final day of each of the three 12-week study periods
  Yes/no

OTHER OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) total symptom score | At the end of the 12-week eplerenone treatment period, compared with the scores at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  Overall summary score between 0 and 100 (0 = very poor health status and 100 = excellent health status)
Six-Minute Walk Test (6MWD) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  Meters walked during six minutes
N-terminal pro b-type natriuretic peptide (NTpro-BNP) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ng/L
eGFR | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  According to the revised Lund-Malmö method in ml/min/1.73 m2
Urine albumine-creatinine ratio | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in mg/mol
Interventricular septal diameter in diastole (IVSd) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in mm, as assessed by TTE
Left ventricular internal diameter in diastole (LVIDd) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in mm, as assessed by TTE
Posterior wall diameter (PWd) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in mm, as assessed by TTE
Left ventricular mass index (LVMi) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in g/m2, as assessed by TTE
Relative wall thickness (RWT) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in %, as assessed by TTE
Stroke volume index (SVI) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ml/m2, as assessed by TTE
Cardiac index (CI) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in l/min/m2, as assessed by TTE
Ejection time | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ms, as assessed by TTE
Indexed left atrial volume (LAVi) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ml/m2, as assessed by TTE
Left atrial (LA) strain | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in %, as assessed by TTE
Indexed left ventricular end diastolic volume (LVEDVi) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ml/m2, as assessed by TTE
Indexed left ventricular end systolic volume (LVESVi) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ml/m2, as assessed by TTE
Left ventricular (LV) EF | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in %, as assessed by TTE
Left ventricular global longitudinal strain (LVGLS) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in %, as assessed by TTE
E/A (early/late ventricular filling velocity) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  ratio, as assessed by TTE
S/D (systolic/diastolic pulmonary vein flow velocity) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  ratio, as assessed by TTE
Isovolumetric contraction velocity (IVCV) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in m/s, as assessed by TTE
Isovolumetric relaxation velocity (IVRV) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in m/s, as assessed by TTE
Isovolumetric relaxation time (IVRT) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ms, as assessed by TTE
Septal S´ | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in cm/s, as assessed by TTE
Lateral S´ | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in cm/s, as assessed by TTE
Septal É | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in cm/s, as assessed by TTE
Lateral É | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in ms, as assessed by TTE
Tricuspid annular plane systolic excursion (TAPSE) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in mm, as assessed by TTE
Right ventricular (RV) strain | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in %, as assessed by TTE
RV S´ | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in cm/s, as assessed by TTE
Systolic pulmonary arterial pressure (SPAP) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in mmHg, as assessed by TTE
Myocardial work index (MWI) | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in mmHg%, as assessed by TTE
Tei index | At the end of the 12-week eplerenone treatment period, compared with the values at the end of the 12-week baseline period and the end of the 12-week withdrawal period
  in %, as assessed by TTE

CONTACTS AND LOCATIONS:
Overall Officials: Krister Lindmark, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Department of Cardiology, Danderyd Hospital, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data with approved ethical permission. All requests will be evaluated, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information will be shared after publication of the results in a peer-reviewed medical journal, and will be available for a minimum of 25 years therafter.
Access Criteria: Access to IPD and supporting information may be granted to qualified researchers whose intended use is to evaluate the trial, provided that participant anonymity is maintained.